CLINICAL TRIAL: NCT05203484
Title: Effect of Multielectrode Versus Point-by-Point Mapping on Recurrence of Ventricular Tachycardia in Ischemic Heart Disease - A Prospective, Randomised Single Centre Trial
Brief Title: Effect of Multielectrode Versus Point-by-Point Mapping on Recurrence of Ventricular Tachycardia in Ischemic Heart Disease
Acronym: EMPIRE-VT
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator left Heart Center Leipzig.
Sponsor: Helios Health Institute GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMPIRE-VT
Record Dates: First submitted 2021-11-29; First posted 2022-01-24 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Ventricular Tachycardia
Keywords: ischemic heart disease; implantable cardioverter-defibrillator; multielectrode mapping; Point-by-Point Mapping
MeSH Terms: conditions — Tachycardia, Ventricular; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multielectrode mapping (Experimental): Participants assigned to the Multielectrode Mapping arm will undergo VT ablation within 48 hours after baseline evaluation. The Mapping procedure will be performed with either a Pentaray or Octaray catheter (Biosense Webster; each 45 catheters, randomly allocated). Catheter ablation of potential diastolic pathways and Scar homogenisation will be performed with a irrigated 3.5mm tip catheter (QDot; Biosense Webster).
  Interventions: Device: Multielecotrde Mapping
- Point-by-Point Mapping (Active Comparator): Participants assigned to the Point-by-Point Mapping arm will undergo VT ablation within 48 hours after baseline evaluation. The Mapping procedure will be performed with a QDot catheter (Biosense Webster). Catheter ablation of potential diastolic pathways and scar homogenisation will also be performed with the QDot catheter.
  Interventions: Device: Point-by-point mapping

INTERVENTIONS:
Device: Multielecotrde Mapping — Multielectrode Mapping with Pentaray/Octaray
  Arms: Multielectrode mapping
Device: Point-by-point mapping — Point-by-point mapping with QDot
  Arms: Point-by-Point Mapping

SUMMARY:
VT ablation is a frequently performed intervention in patients with symptomatic ventricular tachycardia, electrical storm due to monomorphic VT and appropriate ICD shocks, primarily aiming at reducing the burden of complaints, and ICD shocks. The recommendations for its use were described in the ESC guideline for ventricular arrhythmias and the prevention of sudden cardiac death. To visualize the arrhythmogenic substrate leading to ventricular tachycardia complex mapping techniques are currently used in clinical routine, including conventional Point-by-Point mapping or Multielectrode Mapping. The latter is associated with shorter Mapping and overall procedure times, while maintaining the same primary endpoint of the procedure itself. The aim of this trial is to validate, whether the reduction of mapping and procedure time is associated with a comparable long-term outcome compared with conventional Point-by-Point mapping.

DETAILED DESCRIPTION:
Catheter Ablation in Patient with VT and ischemic heart disease has shown a beneficial effect in terms of VT Recurrence and Quality of life. The short-term outcome of catheter Ablation in Patients with this particular disease is good, but VT recurrence during long-term follow up is as high as 50-70%.

An integral Part of the Ablation procedure is the substance guided Mapping for localisation of low Voltage areas, late diastolic or fractioned potentials, as possible substrate for VT maintenance. These diastolic pathways, which represent slow conducting myocardium, are the major prerequisites for Reentry and thus for ventricular tachycardia.

Commonly these diastolic pathways are found in myocardial scar after infarction. Cardiac MRI can help to visualize these scars. In Patients with non-ischemic cardiomyopathy, the physician has to rely on intraprocedural Mapping and localisation of pathologic signals mentioned above.

In the last few years, the use of Multielectrode Mapping catheters becomes more and more part of complex EP procedures, mainly due to a high spatio temporal resolution, thereby reducing the overall Mapping time while maintaining the same primary endpoint of VT-non-inducibility compared to Point-by-Point Mapping.

There is growing evidence, that Multielectrode Mapping is associated with lesser mapping and procedure time, while generating more elecatroanatomical points (and thus more information regarding the arrhythmogenic substrate, responsible for VT maintenance).

Currently there is considerable uncertainty as to whether the reduced mapping and procedure time of Multielectrode Mapping will have an effect on the recurrence of ventricular tachycardia.

Procedure time of catheter ablation in patients with scar mediated ventricular tachycardia is directly correlated to hospital mortality.

Yet there are no prospective studies, which evaluate the effect of the aforementioned Mapping systems in the recurrence of ventricular tachycardia in comparison to conventional mapping techniques.

The objective of the trial is to demonstrate that Multielectrode Mapping in patients with ventricular tachycardia with structural (on inflammatory) is not inferior to conventional Mapping techniques with respect to VT Recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Symptomatic ventricular tachycardia with/without ICD and underlying ischemic
3. No need for coronary revascularisation therapy based on coronary angiography or Cardiac MRI
4. Class I or IIa indication for catheter ablation (according to 2015 Guidelines of the European Society of Cardiology for the management of ventricular tachycardias).
5. Signed informed consent.

Exclusion Criteria:

1. Patients with ventricular assist device
2. Reversible causes of ventricular tachycardia (e. g. thyroid disorder, acute alcohol intoxication, recent major surgical procedures, trauma or acute infection/acute myocarditis)
3. Recent cardiovascular event including myocardial infarction, percutaneous intervention, valve or cardiac bypass surgery
4. Previous VT ablation within the last 3 months
5. Patients with ventricular tachycardia and known atrial fibrillation with sufficient antiarrhythmic drug therapy regarding rhythm control of atrial fibrillation
6. Medical conditions limiting the expected survival to < 1 year
7. On the waiting list for heart transplant.
8. Participation in any other randomized controlled trial
9. Women of childbearing potential without appropriate contraceptive measures (oral contraceptives, vaginal ring, intrauterine devices, implanon, injections, partner with vasectomy)
10. Subjects under legal supervision or guardianship
11. Unable to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
VT recurrence | 12 months
  Time to VT-recurrence based ICD Recordings in dependence of the Mapping modality: Multielectrodemapping with Pentaray/Octaray (Biosense webster) or conventional Point-by-Point mapping with QDOT (Biosense webster)

SECONDARY OUTCOMES:
Comparison of intraprocedural data | directly after procedure
  EAM Points, total mapping and overall procedure time, Mapping quality/accuracy (mapping points used/points acquired), Scar Area, number of RF ablations, RF Ablation time, total fluoroscopy time) in both arms
Rate of ICD shocks/therapies in the follow up period | 12 months
  Total number and date of ATPs/ ICD Shocks, measured by the ICD recordings during the follow up visits
VT Burden | 12 months
  Total number of VT episodes recorded by the ICD in the follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Aarsh Arya, PD, Study Chair — leipzig heart centre; Gerhard Hindricks, Prof. Dr., Study Chair — leipzig heart centre
Locations (1):
- Herzzentrum Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Yes